CLINICAL TRIAL: NCT06295900
Title: The Effect of Aromatherapy Massage Applied to Intensive Care Patients on Sleep Quality
Brief Title: The Effect of Aromatherapy Massage on Sleep Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgün Erdoğan (Other)
Responsible Party: Sponsor-Investigator, Nilgün Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Organization: Nigde Omer Halisdemir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19.10.2023/63
Record Dates: First submitted 2024-01-11; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Respiratory Failure; Pneumonia; Respiratory Disease; Stroke, Ischemic
Keywords: intensive care; sleep quality; aromatherapy massage
MeSH Terms: conditions — Diabetes Mellitus; Respiratory Insufficiency; Pneumonia; Respiration Disorders; Ischemic Stroke; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled single-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 Group (Active Comparator): In this group, application is made with chamomile, lavender and neroli oil.
  Interventions: Other: Intervention 1 Group
- Intervention 2 Group (Sham Comparator): In this group, application is made with lavender oil.
  Interventions: Other: Intervention 2 Group
- Placebo Control Group (Placebo Comparator): In this group, application is made only with almond oil.
  Interventions: Other: Placebo Control Group

INTERVENTIONS:
Other: Intervention 1 Group — 20 patients were included in this group and aromatherapy was applied once a day, for a total of 30 minutes, for three days, with a mixture of lavender, medicinal chamomile, and neroli oil (2 drops of lavender oil, 4 drops of medicinal chamomile, 6 drops of neroli oil in 20 ml of sweet almond oil). Massage is planned.
  Arms: Intervention 1 Group
Other: Intervention 2 Group — It is planned to include 20 patients in this group and perform an aromatherapy massage with a mixture of only lavender oil (12 drops of lavender oil in 20 ml of sweet almond oil), once a day for three days, for a total of 30 minutes.
  Arms: Intervention 2 Group
Other: Placebo Control Group — It is planned to include 20 patients in this group and perform an aromatherapy massage with only almond oil (20 ml sweet almond oil) mixture, once a day for three days, for a total of 30 minutes.
  Arms: Placebo Control Group

SUMMARY:
Sleep disturbance is one of the most common complaints of patients admitted to ICU. Insufficient sleep in intensive care units may be associated with environmental reasons such as excessive light at night, loud warning sounds and mechanical ventilation alarms, as well as non-environmental factors, including the situation at the time of admission. Sleep assessment is subjective in nature, so it is difficult to perform in the ICU. Since communication with the patient is prevented, clear information about perceived rest and disturbing factors cannot be provided. For this reason, night rest is an issue that is often forgotten and ignored. This study applied a mixture of lavender, medicinal chamomile and neroli oil (in 20 ml of sweet almond oil; lavender oil 2 drops, medicinal chamomile 4 drops, neroli oil 6 drops) to patients who were monitored in intensive care on high-flow and oxygen, once a day for three days. This study will be conducted to determine the effect of aromatherapy massage applied for a total of 30 minutes on sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over,
* Conscious patients,
* Staying in intensive care for 24 hours or more,
* Those with stable hemodynamic status,
* Receiving O2 therapy,
* Intubated patients, patients who have passed 24 hours after being extubated,
* Those whose saturation level is 85 and above

Exclusion Criteria:

* Patients with peripheral neuropathy or quadriplegia,
* Patients with open wounds on their body,
* Patients receiving analgesia and sedation infusion,
* Patients who are sedated,
* Patients in delirium,
* Patients with allergies detected before starting the application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient Introduction Form | 1 year
  In the "Patient Introduction Form" prepared by the researcher based on the literature in order to obtain information about the characteristics of the patients who will constitute the sample, the patients' medical diagnosis, age, gender, chronic diseases, length of stay in intensive care, use of analgesic, sedative and hypnotic drugs used, normal sleep hours at night were included. There are questions about (sleep duration, daytime sleep, sleep hours, sleep aids used, etc.).

SECONDARY OUTCOMES:
Patient Follow-up Form | 1 year
  The patient follow-up form was created by the researcher and will include the visual comparison sleep scale follow-up results, the effects of the application (whether side effects develop, its effect on the application area, the patient's condition, etc.) and the dosage of the hypnotic and sedative drugs the patient took in the intensive care unit during the study. The sleep score results of the patients will be recorded on the patient follow-up form by the nurses who collected the data of the study the morning after the application (08), and the effects of the application will also be recorded by the researcher.

OTHER OUTCOMES:
Visual Comparison Sleep Scale | 1 year
  It was first developed by Snyder-Halpern and Verran (1988) in 1987 to evaluate the sleep quality of sick and healthy individuals. The scale consists of 15 questions categorized under three subscales: 'discomfort' (interruptions and delays in sleep), 'effectiveness' (how good sleep rejuvenates the individual) and 'completion' (napping). Disturbance questions include: 1) waking in the middle of sleep, 2) waking after sleep onset, 3) movement during sleep, 4) firmness of sleep, 5) quality of discomfort, 6) sleep latency, and 7) quality of latency. Efficacy questions include: 1) recovery after awakening, 2) subjective sleep quality, 3) sleep adequacy assessment, 4) total sleep time, and 5) total sleep time, calculated by adding total sleep time and waking after sleep onset. Each question is scored using a 100 mm visual analogue scale. For the 'disruption' and 'completion' subscales, higher scores indicate sleep disturbance and lower scores indicate better sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)